CLINICAL TRIAL: NCT06229236
Title: Assessing Effectiveness of a Diabetes Navigator in Increasing Progression (Improving Uptake and/or Optimization) of Advanced Diabetes Technologies
Brief Title: Assessing Effectiveness of a Diabetes Navigator in Increasing Progression of Advanced Diabetes Technologies
Acronym: IMPACT-T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00398788; R01DK134955 (NIH)
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Glucose Monitor (CGM); Insulin Pumps; Hybrid Closed Loop (HCL); Diabetes Navigator; Diabetes Navigator Toolkit; Advanced Diabetes Technology (ADT)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients will be masked until randomization. Outcomes Assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Navigator (Experimental): Support and guidance of Diabetes Navigator in addition to standard care
  Interventions: Behavioral: Diabetes Navigator
- Standard of Care (No Intervention): Standard care provided by the healthcare staff during routine diabetes clinic visits.

INTERVENTIONS:
Behavioral: Diabetes Navigator — Participants in the Diabetes Navigator (DN) arm will receive support from a trained navigator to help them improve progression (improving use/optimization) in use of advanced diabetes technology. The Diabetes Navigator will engage with participants immediately after randomization, throughout the duration of study, using a predefined toolkit, educational resources and interventions to assist them in optimizing use of advanced diabetes technology.
  Arms: Diabetes Navigator

SUMMARY:
The goal of this randomized control trial is to determine if the support of a Diabetes Navigator is more effective than standard care in improving uptake and use of advanced diabetes technology among patients with type 1 diabetes.

DETAILED DESCRIPTION:
This study will recruit 148 individuals, 74 adults (ages 21-75) and 74 youth (ages 5-20) with type 1 diabetes. Participants will be randomized to standard care (usual diabetes care) or the intervention arm in which the participants will receive additional support from a Diabetes Navigator. Participants in the intervention group will receive assistance from a Diabetes Navigator who will help the participants address challenges in acquiring and optimally using advanced diabetes technology. The investigators will compare the group receiving Diabetes Navigator support with the standard care group to see if the additional support improves progression (increases uptake and/or optimization) in use of advanced diabetes technology and, consequently, improves glycemic control among patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 5 to 75 years.
* Diagnosis of type 1 diabetes
* Patient of Johns Hopkins Medicine adult or pediatric diabetes clinics
* Not using or not optimally using diabetes technology.
* Planned Diabetes technology intensification by diabetes provider.
* If already on diabetes technology - must be using the specific device for a minimum of 14 days.

Exclusion Criteria:

* Optimally using Diabetes Technology
* Pregnancy or lactation or planned pregnancy in the next 12 months.
* Other types of diabetes (type 2 diabetes, Maturity Onset Diabetes in Youth, cystic fibrosis-related diabetes, steroid-induced diabetes, post total pancreatectomy, transplant-related diabetes)
* Active participant of any other research study that may interfere with diabetes management.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Percent of participants whose Diabetes Technology Utilization Score (DTUS) increases (based on review of last 14 days of CGM and insulin pump data) | Baseline, 3 months
  Diabetes Technology Utilization Score is calculated based on CGM and Insulin pump use ranging from 0-4, 4 indicating optimal technology use and 0 indicating no use of technology.
  Measured from baseline to 3 months as a binary outcome (yes/no question)

SECONDARY OUTCOMES:
Percent of participants whose Diabetes Technology Utilization Score (DTUS) increases (90 days of data) | Baseline, 3 months
  Diabetes Technology Utilization Score is calculated based on CGM and Insulin pump use ranging from 0-4, 4 indicating optimal technology use and 0 indicating no use of technology. A higher score is better.
  Measured from baseline to 3 months as a binary outcome (yes/no question)
Percent of participants whose Diabetes Technology Utilization Score (DTUS) increases at 3 months and stays the same or increases at 6 months. | Baseline, 3 months, 6 months
  Diabetes Technology Utilization Score is calculated based on CGM and Insulin pump use ranging from 0-4, 4 indicating optimal technology use and 0 indicating no use of technology.
  Measured at 6 months as a binary outcome (yes/no question)
Change in the Diabetes Technology Use Score (DTUS) | Baseline, 3 months and 6 months
  Diabetes Technology Utilization Score is calculated based on CGM and Insulin pump use ranging from 0-4, 4 indicating optimal technology use and 0 indicating no use of technology.
  Measured from baseline to 3 months and from baseline to 6 months. Change measured in difference in points.
Changes in continuous glucose monitor (CGM) "Time in Range" | Baseline, 3 months, 6 months
  Percentage of time blood glucose ranges from 70-180 mg/dL based on CGM data
  Measured as a continuous variable at baseline, 3-months and 6-months.
HbA1c change | Baseline, 3 months, 6 months
  Hemoglobin A1c measured as a continuous variable at baseline, 3-months and 6-months.

OTHER OUTCOMES:
Change in General Technology and Diabetes Technology Attitudes score | Baseline and 6 months
  Measured using General Technology and Diabetes Technology Attitudes survey, a 6-item survey assessing attitudes and use of various general technologies and diabetes devices as reported by participants.
  Min: 1 Max: 5 Mean Score, higher score means better outcome
Change in the Glucose Monitoring Satisfaction Survey score | Baseline and 6 months
  Measured using the Glucose Monitoring Satisfaction Survey (GMSS), a 15-item survey with scores ranging from 0 to 60 with higher scores indicating greater satisfaction.
Change in CGM Benefits and Barriers Scale | Baseline and 6 months
  This survey measures the benefits and burden of Continuous Glucose Monitor (CGM) use as reported by participants.
  Score ranges from 1 (strongly disagree) to 5 (strongly agree). Higher score indicating greater perceived benefits or burdens.
Change in the Diabetes Distress Scale score | Baseline and 6 months
  17 items are scored on a 6-point Likert scale from 1 "not a problem" to 6 "very serious problem." Higher scores mean worse outcome/more distress
Changes in the INSPIRE survey scores | Baseline and 6 months
  The INSPIRE questionnaire assesses user expectations and experiences with Insulin Delivery Systems. Score range 0-100, higher scores indicate a more positive perception of insulin delivery systems. Items are rated on a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree)
Participant reported Acceptability of Intervention Measure (AIM) | 6 months
  Total of 12-items answered on a Likert scale of 1 = completely disagree to 5 = completely agree. Minimum score: 12, maximum score: 60. A higher score indicates greater acceptability of the intervention.
Participant reported Intervention Appropriateness Measure (IAM) | 6 months
  The total score ranges from 4 to 20. Higher scores indicate greater appropriateness.
Participant reported Feasibility of Intervention Measure (FIM) | 6 months
  Feasibility of Intervention Measure includes 4 questions with 5-point likert response options, Completely disagree (1) - Completely agree (5). Higher score, higher agreement of feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Nestoras Mathioudakis, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin T, Manfredo JA, Illesca N, Abiola K, Hwang N, Salsberg S, Akhtar Y, Mathioudakis N, Brown EA, Wolf RM. Improving Continuous Glucose Monitoring Uptake in Underserved Youth with Type 1 Diabetes: The IMPACT Study. Diabetes Technol Ther. 2023 Jan;25(1):13-19. doi: 10.1089/dia.2022.0347. Epub 2022 Nov 7. PMID 36223197
- [Background] Kanbour S, Jones M, Abusamaan MS, Nass C, Everett E, Wolf RM, Sidhaye A, Mathioudakis N. Racial Disparities in Access and Use of Diabetes Technology Among Adult Patients With Type 1 Diabetes in a U.S. Academic Medical Center. Diabetes Care. 2023 Jan 1;46(1):56-64. doi: 10.2337/dc22-1055. PMID 36378855